CLINICAL TRIAL: NCT06836947
Title: The Effect of Two Different Bathing Methods on Vital Signs and Comfort in Pediatric Intensive Care Unit:Bath Trial
Brief Title: The Effect of Two Different Bathing Methods on Vital Signs and Comfort in PICU:Bath Trial
Status: Recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Asst. Prof., Izmir Katip Celebi University
Other Study IDs: 006; ikçü (Other: Katip Çelebi University)
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Vital Sign Monitoring; Comfort
Keywords: pediatrics; bath; nursing care; vital signs; comfort

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional Bathing Group: In traditional bathing, the patient is also bathed in bed with 36-37 degrees water.
- Wipe Bathing Group: Wipe bathing is performed with 36-37 degrees water with 10 ml of chlorhexidine in 200 ml of water.

SUMMARY:
The study was planned to be conducted and completed within 6 months after ethics committee approval was obtained. The study is a prospective, quasi-experimental study.

The population of the study will consist of children who are hospitalized in the Pediatric Intensive Care Unit of SBÜ. İzmir Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital. The vital signs and comfort of the children of the parents who agreed to participate in the study will be measured before bathing (baseline) and care will be taken to ensure that they are similar in both groups.

Children in the study will not be randomized. In the routine operation of the clinic, traditional bathing is performed once a week and wipe bathing is performed once every two days. Wipe bathing is performed at 36-37 degrees water with 10 ml of chlorhexidine in 200 ml of water. Traditional bathing is also performed with 36-37 degrees water in bed or in the bathtub. In the study, no intervention will be performed and the outcomes will be measured and compared with each other before and after both bathing procedures.

Physiologic parameters including respiratory rate, pulse rate, oxygen saturation and comfort levels of newborns just before, during and after the bathing process (1st and 5th minute) will be evaluated and compared with each other. To avoid bias in the study, all bathing procedures will be performed by Specialist Nurse Esat Erdem GÖKPINAR.

Translated with DeepL.com (free version)

DETAILED DESCRIPTION:
The study was planned to be conducted and completed within 6 months after ethics committee approval was obtained. The study is a prospective, quasi-experimental study.

The population of the study will consist of children who are hospitalized in the Pediatric Intensive Care Unit of SBÜ. İzmir Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital. The vital signs and comfort of the children of the parents who agreed to participate in the study will be measured before bathing (baseline) and care will be taken to ensure that they are similar in both groups.

Children in the study will not be randomized. In the routine operation of the clinic, traditional bathing is performed once a week and wipe bathing is performed once every two days. Wipe bathing is performed at 36-37 degrees water with 10 ml of chlorhexidine in 200 ml of water. Traditional bathing is also performed with 36-37 degrees water in bed or in the bathtub. In the study, no intervention will be performed and the outcomes will be measured and compared with each other before and after both bathing procedures.

Physiologic parameters including respiratory rate, pulse rate, oxygen saturation and comfort levels of newborns just before, during and after the bathing process (1st and 5th minute) will be evaluated and compared with each other. To avoid bias in the study, all bathing procedures will be performed by Specialist Nurse Esat Erdem GÖKPINAR.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

1. Being hospitalized in Behçet Uz Pediatric Intensive Care Unit
2. No contraindications to bathing
3. Parent's willingness to participate in the study

Exclusion Criteria:

1. Having a contraindication to bathing
2. Parents were not willing to participate in the study

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: G*power 3.1.9.7 program was used to calculate the sample size required for the study and it was found that a total of 52 patients, 26 patients in each group, should be reached with an effect size of 0.96 (Öz, 2022), power of 0.95 (1-ß) and α:0.05.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Respiration | immediately before and immediately after bath
Pulse | immediately before and immediately after bath
Saturation | immediately before and immediately after bath
Mean Blood pressure | immediately before and immediately after bath
Body Temperature | immediately before and immediately after bath

SECONDARY OUTCOMES:
comfort scale point | immediately before and immediately after bath
  The Comfort scale was developed by Ambuel et al (1992). The Comfort scale is a sedation scoring scale that includes two physiological and six behavioural stress criteria. The sick child is assessed on six behavioural (alertness, calm-agitation, respiratory response, physical movement, muscle tone and facial tension) and two physical parameters (blood pressure and heart rate) within two minutes. Each criterion is scored out of five points. Assessment scores: 27-40: Inadequate sedation, 17-26: Appropriate sedation, 8-16: Excessive sedation. Ambuel et al. reported an internal reliability of 0.84 (p<0.01) for the total score and an internal consistency alpha coefficient of 0.94 for the data collected from 50 observations with 37 patients inthe intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Katip Çelebi University, Cordaleo, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
By ethical rules, patient information will only be shared upon request.